CLINICAL TRIAL: NCT01618071
Title: Unravelling the Mechanisms of Vascular Protection by n3-PUFAs to Optimise and Support Their Use as Bioactives by the Food Industry
Brief Title: Vascular Effects of Triglyceride-rich Lipoproteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Royal Veterinary College (Unknown)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DRINC 11-LO-0116; BB/1005862/1 (Other Grant/Funding Number: BBSRC)
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Postprandial Period; Lipemia; Vasodilation; Vascular Resistance; Nitric Oxide
Keywords: n-3 PUFA; Endothelial cells; Nitric oxide; Oxidative stress; Blood pressure; Vasodilation; Lipemia; Unsaturated dietary fats
MeSH Terms: conditions — Hyperlipidemias; Aneurysm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oleic acid (Active Comparator): 75 g high oleic acid sunflower oil.
  Interventions: Dietary Supplement: High-fat meals varying in their fatty acid composition
- Linoleic acid (Active Comparator): 75 g high linoleic acid sunflower oil.
  Interventions: Dietary Supplement: High-fat meals varying in their fatty acid composition
- Eicosapentaenoic acid and docosahexaenoic acid (Experimental): 5 g EPA and DHA derived from fish oil, made up to a total of 75 g with high oleic sunflower oil.
  Interventions: Dietary Supplement: High-fat meals varying in their fatty acid composition
- Docosahexaenoic acid (Experimental): 5 g DHA derived from algal oil, made up to a total of 75 g with high oleic sunflower oil.
  Interventions: Dietary Supplement: High-fat meals varying in their fatty acid composition

INTERVENTIONS:
Dietary Supplement: High-fat meals varying in their fatty acid composition — 70 g fat incorporated into a muffin and milkshake meal, consumed following fasting baseline measurements
  Other Names: DHASCO; Purified fish oil

SUMMARY:
Many types of cardiovascular disease begin when the layer of cells lining blood vessels (endothelial cells) start to function abnormally. This causes white blood cells (monocytes) to enter the blood vessel wall and eventually form lesions. Fats from foods we consume are carried in the blood for 3-8 hours after a fatty meal in small particles known as chylomicrons (CM) and chylomicron remnants (CMR). The overall aim of this project is to investigate the idea that n-3 polyunsaturated fatty acids (PUFA) protect against heart disease by modifying the effect of CMR on endothelial cells and monocytes. We hypothesize that n3-PUFA carried in CMR reduce detrimental events which promote blood vessel damage and activate protective mechanisms to improve the function of arteries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Non-smokers
* Aged 35-70 years
* Fasting TAG concentrations ≥1.2 mmol/L.

Exclusion Criteria:

* Reported history of CVD (myocardial infarction, angina, venous thrombosis, stroke), impaired fasting glucose/uncontrolled type 2 diabetes (or fasting glucose ≥ 6.1 mmol/L), cancer, kidney, liver or bowel disease.
* Presence of gastrointestinal disorder or use of drug, which is likely to alter gastrointestinal motility or nutrient absorption.
* History of substance abuse or alcoholism (previous weekly alcohol intake >60 units/men)
* Current self-reported weekly alcohol intake exceeding 28 units
* Allergy or intolerance to any component of test meals
* Unwilling to restrict consumption of any source of fish oil for the length of the study
* Weight change of >3kg in preceding 2 months
* Body Mass Index <20 and >35 kg/m2
* Fasting blood cholesterol > 7.8 mmol/L
* Current cigarette smoker.
* Current use of lipid lowering medication

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Activation of inflammatory/oxidative stress pathways within cultured endothelial cells following treatment with 6 h postprandial chylomicron remnant-rich lipoprotein fraction | 6 h post-meal
  The primary outcome of the study is activation of inflammatory/oxidative stress pathways within cultured endothelial cells following incubation with pooled postprandial lipoprotein fractions rich in chylomicron remnants. Due to the nature of this type of research this necessitates more than one primary outcome measure: the primary measures are NF-kappa-beta activation, cytokine production (e.g. interleukin-6) and reactive oxygen species generation in the cultured human endothelial cells.

SECONDARY OUTCOMES:
Incremental area under the plasma concentration versus time curve (iAUC) of triacylglycerol | 0, 1, 2, 3, 4, 5 and 6 h post-meal
Incremental area under the plasma concentration versus time curve (iAUC) of glucose | 0, 1, 2, 3, 4, 5 and 6 h post-meal
Incremental area under the plasma concentration versus time curve (iAUC) for non-esterified fatty acids | 0, 1, 2, 3, 4, 5 and 6 h post-meal
Incremental area under the plasma concentration versus time curve (iAUC) for plasma fatty acid composition (%) | 0, 1, 2, 3, 4, 5 and 6 h post-meal
Incremental area under the plasma concentration versus time curve (iAUC) for cholesterol | 0, 1, 2, 3, 4, 5 and 6 h post-meal
Incremental area under the unit measure versus time curve for brachial augmentation index | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min post-meal
Incremental area under the unit measure versus time curve for systolic blood pressure | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min post-meal
Incremental area under the unit measure versus time curve for diastolic blood pressure | 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 min post-meal
Change in digital volume pulse stiffness index | 0, 2, 4 and 6 h post-meal
Change in digital volume pulse reflection index | 0, 2, 4 and 6 h post-meal
Change in plasma nitrite/nitrate concentrations | 0, 2, 4 and 6 h
Change in plasma 8-isoprostane F2alpha concentrations | 0, 2, 4 and 6 h post-meal
Activation of inflammatory/oxidative stress pathways within cultured endothelial cells following treatment with 4 h postprandial chylomicron remnant-rich lipoprotein fraction | 4 h post-meal
Activation of inflammatory/oxidative stress pathways within cultured endothelial cells following treatment with 5 h postprandial chylomicron remnant-rich lipoprotein fraction | 5 h post-meal

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London, London, United Kingdom

REFERENCES:
- [Background] Lambert MS, Botham KM, Mayes PA. Modification of the fatty acid composition of dietary oils and fats on incorporation into chylomicrons and chylomicron remnants. Br J Nutr. 1996 Sep;76(3):435-45. doi: 10.1079/bjn19960048. PMID 8881715
- [Background] Botham KM, Bravo E, Elliott J, Wheeler-Jones CP. Direct interaction of dietary lipids carried in chylomicron remnants with cells of the artery wall: implications for atherosclerosis development. Curr Pharm Des. 2005;11(28):3681-95. doi: 10.2174/138161205774580732. PMID 16305504
- [Background] Proctor SD, Vine DF, Mamo JC. Arterial retention of apolipoprotein B(48)- and B(100)-containing lipoproteins in atherogenesis. Curr Opin Lipidol. 2002 Oct;13(5):461-70. doi: 10.1097/00041433-200210000-00001. PMID 12352009
- [Background] Marcoux C, Hopkins PN, Wang T, Leary ET, Nakajima K, Davignon J, Cohn JS. Remnant-like particle cholesterol and triglyceride levels of hypertriglyceridemic patients in the fed and fasted state. J Lipid Res. 2000 Sep;41(9):1428-36. PMID 10974050
- [Background] Hall WL, Sanders KA, Sanders TA, Chowienczyk PJ. A high-fat meal enriched with eicosapentaenoic acid reduces postprandial arterial stiffness measured by digital volume pulse analysis in healthy men. J Nutr. 2008 Feb;138(2):287-91. doi: 10.1093/jn/138.2.287. PMID 18203893
- [Background] Burdge GC, Powell J, Dadd T, Talbot D, Civil J, Calder PC. Acute consumption of fish oil improves postprandial VLDL profiles in healthy men aged 50-65 years. Br J Nutr. 2009 Jul;102(1):160-5. doi: 10.1017/S0007114508143550. Epub 2009 Jan 13. PMID 19138437
- [Background] Zampelas A, Peel AS, Gould BJ, Wright J, Williams CM. Polyunsaturated fatty acids of the n-6 and n-3 series: effects on postprandial lipid and apolipoprotein levels in healthy men. Eur J Clin Nutr. 1994 Dec;48(12):842-8. PMID 7889892
- [Background] Armah CK, Jackson KG, Doman I, James L, Cheghani F, Minihane AM. Fish oil fatty acids improve postprandial vascular reactivity in healthy men. Clin Sci (Lond). 2008 Jun;114(11):679-86. doi: 10.1042/CS20070277. PMID 18052925
- [Background] Rontoyanni VG, Hall WL, Pombo-Rodrigues S, Appleton A, Chung R, Sanders TA. A comparison of the changes in cardiac output and systemic vascular resistance during exercise following high-fat meals containing DHA or EPA. Br J Nutr. 2012 Aug;108(3):492-9. doi: 10.1017/S0007114511005721. Epub 2012 Feb 21. PMID 22348439
- [Derived] Purcell R, Latham SH, Botham KM, Hall WL, Wheeler-Jones CP. High-fat meals rich in EPA plus DHA compared with DHA only have differential effects on postprandial lipemia and plasma 8-isoprostane F2alpha concentrations relative to a control high-oleic acid meal: a randomized controlled trial. Am J Clin Nutr. 2014 Oct;100(4):1019-28. doi: 10.3945/ajcn.114.091223. Epub 2014 Aug 6. PMID 25099540
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/25099540